CLINICAL TRIAL: NCT01134536
Title: Open-Label Evaluation of the Pharmacokinetic Profile and Safety of Tapentadol Oral Solution for the Treatment of Postsurgical Pain in Children and Adolescents Aged From 6 to Less Than 18 Years
Brief Title: Pharmacokinetics and Safety Study of Tapentadol for Postsurgical Pain in Children and Adolescents
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Collaborators: Grünenthal GmbH (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR016891; R331333PAI2005 (Other: Janssen Research & Development, LLC); KF59 (Other: Janssen Research & Development, LLC); 2010-020380-20 (Other: Janssen Research & Development, LLC); KF5503/59 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2010-05-28; First posted 2010-06-02 (Estimated); Last update posted 2014-07-14 (Estimated); Status verified 2014-07

CONDITIONS: Pain, Postoperative; Postoperative Pain
Keywords: Pain, Postoperative; Postoperative Pain; Tapentadol; NUCYNTA; CG5503; R331333; Pharmacokinetics; Postsurgical pain; Children; Adolescents
MeSH Terms: conditions — Pain, Postoperative | interventions — Tapentadol; Solutions

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Tapentadol Oral Solution (OS) (Experimental)
  Interventions: Drug: Tapentadol (OS) Oral Solution

INTERVENTIONS:
Drug: Tapentadol (OS) Oral Solution — Tapentadol OS Bodyweight <20 kg: Type=4 unit=mg/mL form=oral solution route=oral use or Tapentadol OS Bodyweight >=20 kg: Type=20 unit=mg/mL form=oral solution route=oral use. Single oral dose administered once.

SUMMARY:
The purpose of this study is to evaluate the pharmacokinetic (PK) profile; and safety and tolerability of a single dose of tapentadol oral solution (OS) 1 mg/kg in children and adolescents aged from 6 to less than 18 years with acute, moderate to severe postsurgical pain.

DETAILED DESCRIPTION:
This is a multicenter, single-arm, open-label (all people involved know the identity of the intervention), single-dose study to evaluate the pharmacokinetic (PK) profile (how drugs are absorbed in the body, how they are distributed within the body and how they are removed from the body over time), safety and tolerability of tapentadol 1 mg/kg oral solution (OS) in children aged from 6 to less than 18 years after scheduled surgical procedures that routinely produce acute, moderate to severe postsurgical pain. A screening phase, as per standard of care but not exceeding 30 days, will include the preoperative evaluation, the surgical procedure and its immediate post recovery, and will be followed by the open-label treatment phase and end-of-study assessments. Study drug administration will take place after the surgery has been completed, when the patient is alert, orientated, able to follow commands and complete the required postoperative procedures, and able to tolerate fluid and medication orally. Confinement to the study center for a patient will be as per standard of care, and will include the surgery, the entire 15-hour postdose evaluation period and the end-of-study evaluations. Children with a body weight less than 20 kg will be dosed with a single dose of tapentadol 4 mg/mL OS and children with a body weight of 20 kg or greater will be dosed with a single dose of tapentadol 20 mg/mL OS.

ELIGIBILITY:
Inclusion Criteria:

* Parent(s) or the legal guardian(s) of the patient signed an informed consent document indicating that they understand the purpose of the study, the risks and benefits of the procedures required for the study and give permission for their child to participate in the study
* Physical status rated as I or II on the American Society of Anesthesiologists (ASA) rating scale
* Patient is alert, oriented, able to follow commands, able to understand the study requirements and procedures, and able to communicate intelligibly with the health care provider (taking into account his/her age)
* As per investigator's medical evaluation, patient is able to drink and tolerate oral fluids and medication
* Patient has a postoperative pain intensity score >=4 on the McGrath Color Analog Scale (CAS) as a result of a scheduled surgical procedure or if in the investigator's clinical judgment (ie, investigator judgment relying on standard of care rather than the McGrath CAS), the patient has a pain level that the standard of care following the surgical procedure (which reliably produces moderate to severe pain) requires opioid treatment

Exclusion Criteria:

* History of seizure disorder or epilepsy, or serotonin syndrome, or mild or moderate traumatic brain injury, stroke, transient ischemic attack, or brain neoplasm within 1 year of screening, or severe traumatic brain injury within 15 years of screening, or any traumatic or hypoxic brain injury resulting in ongoing sequelae suggesting transient changes in consciousness
* Moderate to severe renal or hepatic impairment
* Requires concomitant use of sedatives, other than those used during surgery
* Has received dextromethorphan within 2 days before the scheduled study drug administration.

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 45 (Actual)
Dates: Start 2011-10; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic profile | 15 hours after the dose

SECONDARY OUTCOMES:
number of patients with adverse events as a measure of safety and tolerability | end of treatment (from 15 hours post treatment to discharge or early withdrawal)
Number of patients with adverse events as a measure of safety and tolerability | Up to 15 hours post treatment on Day 1

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC C. Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (17):
- United States (10):
  - Little Rock, Arkansas
  - Washington D.C., District of Columbia
  - Meridian, Idaho
  - Ann Arbor, Michigan
  - The Bronx, New York
  - Charlotte, North Carolina
  - Durham, North Carolina
  - Toledo, Ohio
  - Pittsburgh, Pennsylvania
  - Salt Lake City, Utah
- Canada (3):
  - Hamilton, Ontario
  - Ottawa, Ontario
  - Sherbrooke, Quebec
- France (2):
  - F-75 730 Paris Cedex 15
  - Rennes
- Spain (2):
  - Madrid
  - Valladolid

REFERENCES:
- See also: Open-Label Evaluation of the Pharmacokinetic Profile and Safety of Tapentadol Oral Solution for the Treatment of Postsurgical Pain in Children and Adolescents Aged From 6 to Less Than 18 Years — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=837&filename=CR016891_CSR.pdf